CLINICAL TRIAL: NCT00148993
Title: Allogeneic Tumor Cell Vaccination in Patients With Solid Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI (Prof. Slavin) not longer work at Hadassah
Sponsor: Hadassah Medical Organization (Other)
Collaborators: The International Center for Cell Therapy & Cancer Immunotherapy (CTCI) (Unknown)
Responsible Party: Shimon Slavin MD, The International Center for Cell Therapy & Cancer Immunotherapy (CTCI)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 100798-HMO-CTIL
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2005-07

CONDITIONS: Metastatic Solid Tumors
Keywords: Tumor cell vaccine
MeSH Terms: interventions — FANG vaccine

INTERVENTIONS:
Biological: Tumor Cell Vaccine

SUMMARY:
The goal of this study is to apply allogeneic tumor cell vaccination for immunotherapy in patients with micro-metastatic disease and/or in patients at high risk disease progression. The present study will use allogeneic tumor cell lines for tumor cell vaccines that share MHC determinants with the patient aiming to overcome possible restriction of antigen presentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable metastatic disease or disease resistant to chemotherapy or with minimal residual disease at high risk to relapse.

Exclusion Criteria:

* Karnofsky less than 60%. Unrelated condition requiring the use of any cytotoxic agents or immunosuppressive agents which may interfere with optimal immune response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 1998-07; Study Completion 2005-07 (Estimated)

PRIMARY OUTCOMES:
Investigate the feasibility of anti-tumor immune response by allogeneic tumor cell vaccine using tumor cells that share MHC determinants with the patient.

SECONDARY OUTCOMES:
Investigate the feasibility of immune responses against cancer cells by combining allogeneic TCV with indomethacin, cimetidine, tetanus and rIL-2.

CONTACTS AND LOCATIONS:
Overall Officials: shimon slavin, MD, Principal Investigator — The International Center for Cell Therapy & Cancer Immunotherapy (CTCI)
Locations (1):
- The International Center for Cell Therapy & Cancer Immunotherapy (CTCI), Tel Aviv, Israel